CLINICAL TRIAL: NCT01613131
Title: Effectiveness of Perimenopausal Hormone Therapy in Suppression of Ovulation, Stabilization of Reproductive Hormones and Symptom Control
Brief Title: Mirena and Estrogen for Control of Perimenopause Symptoms and Ovulation Suppression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-1711
Record Dates: First submitted 2012-06-04; First posted 2012-06-06 (Estimated); Results first posted 2015-12-02 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-10

CONDITIONS: Menopausal and Other Perimenopausal Disorders
MeSH Terms: interventions — Levonorgestrel; Estradiol; Dichlorodiphenyldichloroethane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mirena + Estradiol Gel (Active Comparator): Subjects will be assigned to use of Estradiol gel for use with Mirena.
  Interventions: Drug: Mirena; Drug: Estradiol
- Mirena + Placebo Gel (Placebo Comparator): Subjects will be assigned to use of placebo gel for use with Mirena.
  Interventions: Drug: Mirena; Drug: Placebo Gel

INTERVENTIONS:
Drug: Mirena — Mirena (levonorgestrel-releasing intrauterine system), 52 mg (20 mcg/day), 5 year duration (study duration 6 months).
  Other Names: IUD
Drug: Estradiol — Topical, .06%, Applied once daily for 50 days.
  Other Names: TDE
  Arms: Mirena + Estradiol Gel
Drug: Placebo Gel — Topical Gel, Applied once daily for 50 days, Placebo comparator.
  Other Names: placebo
  Arms: Mirena + Placebo Gel

SUMMARY:
Hormonal treatment of perimenopausal women has frequently utilized oral contraceptive pills (OCPs). Because of their ability to suppress ovulation and establish cycle control, OCPs have become a popular option, and one that is FDA approved for use until menopause. However, use of OCPs in women in their 40's and 50's carries significant cardiovascular risks. Venous thromboembolism risk is 3-6 fold greater in OCP users, and the risk of myocardial infarction (MI) is approximately doubled in OCP users over the age of 40. This occurs at an age where the background population risk of MI begins to increase, such that the absolute number of cases rises substantially. Women with additional risk factors for cardiovascular disease have a much greater risk for MI (6-40-fold) in association with OCPs. There are also large subgroups of midlife women who are not candidates for OCP use, such a smokers and migraineurs. Moreover, the trend towards lower estrogen dosing with OCPs containing 20 micrograms of ethinyl estradiol has not led to a detectable decrease in thromboembolic risk.

Because of their increased potential risks, it is appropriate to seek alternatives to OCPs and to explore lower doses of hormones to relieve perimenopausal symptoms that occur prior to a woman's final menses. Recent evidence indicates that the hypothalamic-pituitary axis of reproductively aging women is more susceptible to suppression by sex steroids that previously believed. It is possible that hormone doses as low as 50 micrograms of transdermal estradiol (TDE) can suppress the hypothalamic-pituitary axis of midlife women. It is also tempting to speculate that the low but measurable circulating doses of levonorgestrel that are present when a woman uses the Mirena intrauterine system (IUS) can contribute to or even independently suppress the hypothalamic-pituitary axis, and reduce the hormonal fluctuations that result in worsening of perimenopausal symptoms. The combination of low dose TDE plus Mirena may therefore confer superior symptom control as well as contraceptive effectiveness, at far less risk.

DETAILED DESCRIPTION:
The Specific Aims of the present proposal are therefore as follows:

Aim 1: To test the hypothesis that low dose estrogen therapy in concert with the low doses of levonorgestrel that circulate when Mirena is used will suppress ovulation in perimenopausal women.

Aim 2: To examine ovulation rates and symptom control with Mirena alone, and to assess the tolerability of combined estrogen therapy plus the Mirena IUS as a treatment option for symptomatic perimenopausal women.

The proposed pilot study is designed to test the feasibility and tolerability of the proposed regimens: Mirena alone or Mirena plus low-dose TDE in treating symptoms in perimenopausal women and to provide the preliminary data for a larger, comparative effectiveness study of optimal symptom control and provision of long term contraception for midlife women within 5 years of their final menstrual period.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-52
* History of regular menstrual cycles every 20-35 days in mid-reproductive life (20-35 years of age)
* At least 1 period within the past 3 months
* BMI less than 35 kg/m2
* Presence of at least one of the following perimenopausal symptoms:

  1. Hot flashes (vasomotor symptoms)
  2. Cyclical headache, bloating or adverse mood
  3. Self-reported poor quality of sleep

Exclusion Criteria:

* Age < 40 years
* Hysterectomy or bilateral oophorectomy
* Cigarette smoking
* Signs or symptoms of restless leg syndrome or sleep apnea
* Any chronic renal or hepatic disease that might interfere with excretion of gonadotropins or sex steroids
* Moderate/vigorous aerobic exercise > 4 hours per week
* Inability to read/write English
* Pregnant Women
* Prisoners
* Decisionally challenged subjects
* Any medical condition that makes use of Topical estradiol or Mirena contraindicated.
* Sex hormone use within the past 30 days
* History of cancer, blood clots or blood clotting disorder

Ages: 40 Years to 52 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2012-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nanette Santoro, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women were recruited from the University of Colorado Denver campus by direct physician referral or from advertisements in the University community.
Pre-assignment Details: Women using systemic hormonal contraception (patch, pill, ring) were required to have a 30 day hormone washout prior to placement. One subject signed the consent, but failed to meet the inclusion/exclusion criteria during the screening process. Thus, there were 39 women that were enrolled, but only 38 that started in the participant flow.
Period: Overall Study
Arm/Group | Mirena + Estradiol Gel | Mirena + Placebo Gel
Started | 20 | 18
Completed | 17 | 13
Not Completed | 3 | 5
Not completed — Withdrawal by Subject | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mirena + Estradiol Gel | Mirena + Placebo Gel | Total
Number analyzed (Participants) | 20 | 18 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 18 | 38
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 38
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 18 | 38

OUTCOME MEASURES:

1. Primary Outcome: Hot Flashes
Description: The Hot Flash Related Daily Interference Scale (HFRDIS) is a ten item scale measuring degree to which hot flashes interfere with 9 daily activities (work, social, leisure, sleep, mood, concentration, relations, sexuality, enjoyment of life, overall quality of life) over the prior week, each scored on a 10 point Likert scale. The total score is reported, and scores range from 0-100, 100 being the worst outcome.
Time Frame: Day 0
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Mirena + Estradiol Gel | Mirena + Placebo Gel
Number analyzed (Participants) | 20 | 18
scores on a scale | 10.3 (2.653) | 7.944 (2.85)

2. Primary Outcome: Sleep
Description: The Pittsburgh Sleep Quality Index (PSQI) is a 19-item scale designed to measure general sleep disturbances over the previous month (sleep wake patterns, duration of sleep, sleep latency, impact of poor sleep on daytime functioning, assesses specific problems contributing to poor sleep, including pain, urination, breathing difficulty, snoring, dreams, temperature). The global score is reported and ranges from 1-21, with higher scores being indicative of poorer sleep.
Time Frame: Day 0
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Mirena + Estradiol Gel | Mirena + Placebo Gel
Number analyzed (Participants) | 20 | 18
scores on a scale | 9.80 (1.13) | 8.83 (1.01)

3. Primary Outcome: Depression
Description: The Center for Epidemiologic Studies-Depression Scale (CES-D) is a 20-item scale with 4-point Likert responses indicating frequency of symptoms over past week. Scores range from 0-60, with scores >16 considered indicative of depressive symptoms.
Time Frame: Day 0
Population: Two women in the Mirena + Placebo Gel did not provide complete data for this outcome measure; thus they were not included in the analysis for this timepoint.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Mirena + Estradiol Gel | Mirena + Placebo Gel
Number analyzed (Participants) | 20 | 16
scores on a scale | 9.8 (1.34) | 11.31 (2.27)

4. Primary Outcome: Fatigue
Description: The Fatigue Severity Scale (FSS) was used to determine the degree to which night-time sleep difficulty manifested as daytime sleepiness. The FSS is a 9-item scale assessing fatigue over the past week, on a 7-point Likert scale (ranging from 1-7). It is scored by averaging the individual item scores, with higher scores indicating greater fatigue. Scores greater than or equal to 5.5 are generally indicative of insomnia with impaired daytime functioning.
Time Frame: Day 0
Population: One woman in the Mirena + Placebo Gel arm did not provide complete data for this outcome measure; thus she was not included in the analysis for this timepoint.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Mirena + Estradiol Gel | Mirena + Placebo Gel
Number analyzed (Participants) | 20 | 17
scores on a scale | 3.38 (.32) | 3.90 (.34)

5. Primary Outcome: Sleep
Description: as for outcome 2
Time Frame: Day 90
Population: 3 women in the Mirena + Estradiol Gel arm, and 5 women in the Mirena + Placebo Gel did not provide complete data; thus, were not included in the analysis for this timepoint.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Mirena + Estradiol Gel | Mirena + Placebo Gel
Number analyzed (Participants) | 17 | 13
scores on a scale | 9.24 (1.04) | 9.31 (1.37)

6. Primary Outcome: Sleep
Description: as for outcome 2
Time Frame: Day 140
Population: 5 women in the Mirena + Estradiol Gel arm, and 7 women in the Mirena + Placebo Gel did not provide complete data; thus, were not included in the analysis for this timepoint.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Mirena + Estradiol Gel | Mirena + Placebo Gel
Number analyzed (Participants) | 15 | 11
scores on a scale | 8.67 (1.10) | 7.46 (1.46)

7. Primary Outcome: Hot Flashes
Description: as for outcome 1
Time Frame: Day 90
Population: as for outcome 5
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Mirena + Estradiol Gel | Mirena + Placebo Gel
Number analyzed (Participants) | 17 | 13
scores on a scale | 12.71 (3.70) | 5.31 (2.62)

8. Primary Outcome: Hot Flashes
Description: as for outcome 1
Time Frame: Day 140
Population: 3 women in the Mirena + Estradiol Gel arm, and 5 women in the Mirena + Placebo Gel did not provide data; thus, were not included in the analysis for this timepoint.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Mirena + Estradiol Gel | Mirena + Placebo Gel
Number analyzed (Participants) | 17 | 13
scores on a scale | 7.18 (2.12) | 9.54 (4.09)

9. Primary Outcome: Depression
Description: as for outcome 3
Time Frame: Day 90
Population: 4 women in the Mirena + Estradiol Gel arm, and 5 women in the Mirena + Placebo Gel did not provide complete data; thus, were not included in the analysis for this timepoint.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Mirena + Estradiol Gel | Mirena + Placebo Gel
Number analyzed (Participants) | 16 | 13
scores on a scale | 9.69 (1.46) | 11.46 (2.92)

10. Primary Outcome: Depression
Description: as for outcome 3
Time Frame: Day 140
Population: 3 women in the Mirena + Estradiol Gel arm, and 6 women in the Mirena + Placebo Gel did not provide complete data; thus, were not included in the analysis for this timepoint.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Mirena + Estradiol Gel | Mirena + Placebo Gel
Number analyzed (Participants) | 17 | 12
scores on a scale | 11.41 (1.80) | 12.08 (2.56)

11. Primary Outcome: Fatigue
Description: as for outcome 4
Time Frame: Day 90
Population: as for outcome 10
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Mirena + Estradiol Gel | Mirena + Placebo Gel
Number analyzed (Participants) | 17 | 12
scores on a scale | 3.54 (.34) | 3.80 (.35)

12. Primary Outcome: Fatigue
Description: as for outcome 4
Time Frame: Day 140
Population: as for outcome 5
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Mirena + Estradiol Gel | Mirena + Placebo Gel
Number analyzed (Participants) | 17 | 13
scores on a scale | 2.78 (.27) | 3.90 (.39)

ADVERSE EVENTS:
Time Frame: 140 days
Arm/Group | Mirena + Estradiol Gel | Mirena + Placebo Gel
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/18
Other Adverse Events (participants affected / at risk) | 1/20 | 1/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirena + Estradiol Gel (N=20) | Mirena + Placebo Gel (N=18)
Mood changes (General disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
The main limitation was the sample size, which is consistent with a pilot study, and which can only inform the design of future research.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No